CLINICAL TRIAL: NCT05481580
Title: Relationship Between Molar Restoration and Furcation Involvement
Brief Title: Restorations and Furcation Involvement on Molars
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Nicola Alberto Valente, DDS, MS, PhD, Assistant Professor, University of Cagliari
Other Study IDs: Perio2
Record Dates: First submitted 2022-07-25; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Furcation Defects
Keywords: Furcation Defects; Dental Restoration, Permanent; Dental Crowns
MeSH Terms: conditions — Furcation Defects | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Restored: Molars with a 2nd class restoration or a crown
  Interventions: Diagnostic Test: Periodontal probing
- Non-restored: Molars with no restorations
  Interventions: Diagnostic Test: Periodontal probing

INTERVENTIONS:
Diagnostic Test: Periodontal probing — The teeth involved will be probed to assess probing depth, presence of furcation, bleeding.
  A radiograph will be taken to assess the length of the root trunk and the presence of root canal treatment
  Other Names: Radiograph

SUMMARY:
The aim of this study will be to analyze the relationship between the presence of second class restorations (interproximal fillings) or prostheses (crowns, bridges) on molar teeth and the presence of bone resorption between the roots of the latter. Patients with this type of restorations will be identified and a non-interventional clinical and radiographic analysis will be conducted.

DETAILED DESCRIPTION:
Patients who have a molar tooth reconstructed with a second class filling according to Black, or a with crown or that is abutment of a prosthetic bridge will be included in the study provided they have at least one other intact molar.

The molars included in the study do not have to be wisdom teeth. In these patients, in addition to the presence of furcations (bone resorption in the space between the roots), the probing depth (PD), the loss of clinical attachment (CAL), bleeding on probing ( BOP), mobility, width of the keratinized tissue, the length of the root trunk (measured radiographically), the presence or absence of endodontic treatments (evaluated on the radiography), the anatomy of the roots (widely separated, fused, separated but fused) and the presence of enamel projections will be recorded.

Data will be analyzed with utilizing Pearson chi-square and the pair-wise t test.

The analysis of these data will provide us with evidence on the influence that interproximal restorations and fixed prostheses, in the presence of other co-factors, have on the presence of furcations in molars.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have molars both with and without restorations
* Restorations presents for at least 5 years

Exclusion Criteria:

* Patients who do not want to undergo evaluation
* Patients who cannot undergo radiation (pregnant women)
* Patients who do not have at least one other unrestored molar

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Periodontal maintenance patients who have restored and non-restored molars present both with and without furcation involvement.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Presence of furcation | At the time of evaluation, the first time the patients is seen (time 0)
  The presence of bone resorption between the roots of the molar

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Duilio Casula, AOU Cagliari, Monserrato, CA, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared in a publication after the end of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be submitted for publication right after the analysis of the outcomes

REFERENCES:
- [Background] Nibali L, Zavattini A, Nagata K, Di Iorio A, Lin GH, Needleman I, Donos N. Tooth loss in molars with and without furcation involvement - a systematic review and meta-analysis. J Clin Periodontol. 2016 Feb;43(2):156-66. doi: 10.1111/jcpe.12497. Epub 2016 Feb 12. PMID 26932323
- [Result] Wang HL, Burgett FG, Shyr Y. The relationship between restoration and furcation involvement on molar teeth. J Periodontol. 1993 Apr;64(4):302-5. doi: 10.1902/jop.1993.64.4.302. PMID 8483093
- [Result] Hou GL, Tsai CC. Relationship between periodontal furcation involvement and molar cervical enamel projections. J Periodontol. 1987 Oct;58(10):715-21. doi: 10.1902/jop.1987.58.10.715. PMID 3478466
- [Result] Brunsvold MA, Lane JJ. The prevalence of overhanging dental restorations and their relationship to periodontal disease. J Clin Periodontol. 1990 Feb;17(2):67-72. doi: 10.1111/j.1600-051x.1990.tb01064.x. PMID 2406294